CLINICAL TRIAL: NCT07367022
Title: The Accuracy of Portable Sleep Monitoring for Children With Autism Spectrum Disorder
Brief Title: Portable Sleep Monitors in Children With Autism Spectrum Disorder
Acronym: PrSM
Status: Recruiting | Type: Observational
Sponsor: Lena Xiao (Other)
Responsible Party: Sponsor-Investigator, Lena Xiao, Clinical Assistant Professor, University of British Columbia
Organization: University of British Columbia (Other)
Other Study IDs: H25-00532
Record Dates: First submitted 2025-09-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder (ASD); Obstructive Sleep Apnea (OSA)
Keywords: Portable Sleep Monitor; Polysomnogram; Children with ASD; Nox T3s; Sleep Disordered Breathing; Sleep disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with ASD testing a portable sleep monitor: Children aged 6-18 years old with autism spectrum disorder concurrently testing a portable sleep monitor (Nox T3s) during their first clinical polysomnogram. Children and their caregivers may also complete a qualitative interview about sleep testing preferences after their sleep test.
  Interventions: Device: Portable sleep monitor (Nox T3s)

INTERVENTIONS:
Device: Portable sleep monitor (Nox T3s) — Participants will test the Nox T3s portable sleep monitor concurrently during their in-hospital clinical polysomnogram.

SUMMARY:
The goal of this study is to evaluate the ability of a portable sleep monitor to detect obstructive sleep apnea in children with autism spectrum disorder (ASD). The main study objectives are to:

1. Evaluate the correlation between the obstructive apnea-hypopnea index (OAHI) on a portable sleep monitor and an in-laboratory polysomnogram (PSG);
2. Determine the sensitivity and specificity of a portable sleep monitor to diagnose obstructive sleep apnea (OSA);
3. Evaluate patient and family preferences for sleep testing.

DETAILED DESCRIPTION:
Sleep disorders are highly prevalent in children with ASD, with as many as 80% of children reporting poor sleep. To identify the cause of poor sleep, many children will require a sleep study (polysomnogram; PSG), which is an overnight study done at the hospital using many different sensors to measure sleep and breathing. The PSG is the gold standard diagnostic test for obstructive sleep apnea (OSA) and measures the rate of obstructive respiratory events during sleep (obstructive apnea-hypopnea index; OAHI) which is crucial for treatment decision-making. However, PSGs are challenging for children with ASD due to the disrupted routine, burden and stress, and intolerance to the PSG setup. Further, diagnosis may be delayed up to 2 years due to a lack of pediatric sleep facilities in Canada, with pronounced geographical disparities. Although sleep disturbances are prevalent amongst children with ASD, there are significant inequities in accessing pediatric sleep medicine care and diagnostic testing. Alternative, simpler diagnostic testing is needed.

We will evaluate a portable sleep monitor as the first step towards establishing home sleep apnea testing in children with ASD. We will conduct a feasibility study testing the Nox T3s portable sleep monitor alongside the traditional in-hospital polysomnogram to compare the ability of the Nox T3s to identify obstructive sleep apnea in children with ASD. We will also conduct qualitative interviews with families to gather insight on participant and family preferences for sleep testing to better address the needs of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 6 to 18 years of age, AND;
2. Children diagnosed with autism spectrum disorder, AND;
3. Children who will be undergoing a polysomnogram (PSG) for the first time, AND;
4. Caregiver willing to complete questionnaires about child's sleep and behavior

Exclusion Criteria:

1. Children who are currently using respiratory therapy
2. Children who have previously completed a PSG
3. Caregiver unwilling to complete questionnaires about child's sleep and behavior

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who are undergoing a clinical PSG at British Columbia's Children's Hospital in Vancouver, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Obstructive Apnea-Hypopnea Index (OAHI) measured from the portable sleep monitor and from the polysomnogram (PSG) | Baseline
  The OAHI measured from the portable sleep monitor will be compared to the OAHI measured from the PSG, the gold standard test for sleep-disordered breathing, to determine the ability of the portable sleep monitor to diagnose obstructive sleep apnea.

SECONDARY OUTCOMES:
Patient and Family Preferences | 0-3 months after the baseline PSG
  Optional semi-structured qualitative interviews with caregivers and the patient, if they choose to and are capable of participating in the interviews. The interviews will be conducted virtually by a study team member to explore patient and family preferences and experiences with diagnostic sleep testing.
Insomnia Questionnaire | +/- 1 week from baseline PSG sleep test
  The caregiver-reported Pediatric Insomnia Severity Index will be used to measure the severity of pediatric insomnia symptoms. Scores range from 0 to 30, with higher scores indicating greater insomnia severity.
Chronotype Questionnaire | +/- 1 week from baseline PSG sleep test
  The caregiver-reported Children's Chronotype Questionnaire will measure the chronotype of the participant. The caregiver is given a short description of different chronotypes and selects the chronotype that best reflects their child's preference from a 5-point scale, ranging from "Definitely a Morning Type" = 1 to "Definitely an Evening Type" = 5.
Chronotype Questionnaire | +/- 1 week from baseline PSG sleep test
  The Morningness/Eveningness Scale from the caregiver-reported Children's Chronotype Questionnaire will measure the participant's differences in activeness and alertness in the mornings and evenings. Scores range from 10-48, with scores indicating a morning type (≤ 23), intermediate type (24-32), and evening type (≥33).
Chronotype Questionnaire | +/- 1 week from baseline PSG sleep test
  The sleep and wake parameters from the caregiver-reported Children's Chronotype Questionnaire will measure the participant's midsleep point on free days (MSF).
Sleep Questionnaire | +/- 1 week from baseline PSG sleep test
  The caregiver-reported Pediatric Sleep Questionnaire: Sleep-Related Breathing Disorders subscale will measure the risk for sleep-related breathing disorders. The questionnaire contains 22-items scored as "yes" = 1 and "no" = 0 and normalized to the total number of questions answered, yielding a score between 0.0-1.0. Scores >0.33 indicate a high risk for sleep-related breathing disorders.
Psychological Scale (Emotional Symptoms) | +/- 1 week from baseline PSG sleep test
  The Emotional Symptoms subscale of the Strengths and Difficulties Questionnaire will be used. The 5-item subscale score ranges from 0-10, with greater scores indicating greater emotional difficulties.
Psychological Scale (Conduct Problems) | +/- 1 week from baseline PSG sleep test
  The Conduct Problems subscale of the Strengths and Difficulties Questionnaire will be used. The 5-item subscale score ranges from 0-10, with greater scores indicating greater conduct difficulties.
Psychological Scale (Hyperactivity/inattention) | +/- 1 week from baseline PSG sleep test
  The Hyperactivity/inattention subscale of the Strengths and Difficulties Questionnaire will be used. The 5-item subscale score ranges from 0-10, with greater scores indicating greater hyperactivity/inattention problems.
Psychological Scale (Peer Relationship Problems) | +/- 1 week from baseline PSG sleep test
  The Peer Relationship Problems subscale of the Strengths and Difficulties Questionnaire will be used. The 5-item subscale score ranges from 0-10, with greater scores indicating greater peer relationship problems.
Psychological Scale (Pro-Social) | +/- 1 week from baseline PSG sleep test
  The Pro-Social subscale of the Strengths and Difficulties Questionnaire will be used. The 5-item subscale score ranges from 0-10, with greater scores indicating less difficulty and an increased aptitude for kind and helpful behaviour.
Psychological Scale (Total Difficulties) | +/- 1 week from baseline PSG sleep test
  The Total Difficulties/Overall Stress scale of the Strengths and Difficulties Questionnaire will be calculated by totaling the following 4 subscales: emotional, conduct, hyperactivity, and peer relationships. The total score ranges from 0-40, with greater scores indicating greater difficulties and overall stress.
Sensory Scale (Auditory Hypersensitivity) | +/- 1 week from baseline PSG sleep test
  The Auditory Hypersensitivity subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 9-36, with greater scores indicating higher sensitivity for, and problems with, sounds related to auditory danger signals.
Sensory Scale (Auditory Hyposensitivity to Voices) | +/- 1 week from baseline PSG sleep test
  The Auditory Hyposensitivity to Voices subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 5-20, with greater scores indicating reduced sensitivity for speech or voices.
Sensory Scale (Visual Hypersensitivity) | +/- 1 week from baseline PSG sleep test
  The Visual Hypersensitivity subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 10-40, with greater scores indicating increased sensitivity to light and movement.
Sensory Scale (Tactile Hypersensitivity) | +/- 1 week from baseline PSG sleep test
  The Tactile Hypersensitivity subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 10-40, with greater scores indicating increased sensitivity to non-social touch.
Sensory Scale (Affiliative Touch Aversion) | +/- 1 week from baseline PSG sleep test
  The Affiliative Touch Aversion subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 3-12, with greater scores indicating increased negative response to social touch.
Sensory Scale (Selective Eating) | +/- 1 week from baseline PSG sleep test
  The Selective Eating subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 6-24, with greater scores indicating increased selectivity in food choices (i.e. picky eating).
Sensory Scale (Ingestive Problems) | +/- 1 week from baseline PSG sleep test
  The Ingestive Problems subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 3-12, with greater scores indicating increased problems with swallowing and retaining food.
Sensory Scale (Digestive Problems) | +/- 1 week from baseline PSG sleep test
  The Digestive Problems subscale of the Body Brain Center Sensory Scales will be used. The subscale score ranges from 4-16, with greater scores indicating increased problems with digestion.
Autism Symptoms Dimensions Scale | +/- 1 week from baseline PSG sleep test
  The caregiver-reported Autism Symptoms Dimensions Scale (ASDS) will be used to measure core autism symptoms in children and adolescents. The 39-item questionnaire is scored on a 5-point scale with total ASDS scores ranging from 39-195. Scores between 114-130 indicate high symptom levels and scores >130 indicate very high symptom levels.

CONTACTS AND LOCATIONS:
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided